CLINICAL TRIAL: NCT03122730
Title: A Two-Part Pharmacodynamic Study to Compare VentaProst (Epoprostenol Solution for Inhalation Via Custom Drug Delivery System) Dosing to Conventionally Administered Aerosolized Epoprostenol Dosing in Cardiac Surgery Patients
Brief Title: VentaProst Versus Conventionally-Administered Aerosolized Epoprostenol in Patients Undergoing Cardiac Surgery With CPB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerogen Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APC-VP-CLN-001
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension
Keywords: Cardiac surgery; Cardiopulmonary bypass; Epoprostenol
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VentaProst (Experimental): VentaProst (epoprostenol solution for inhalation via custom drug delivery system)
  In Part 1, subjects were treated with a commercial aerosolized epoprostenol and then removed from that treatment. VentaProst was started and titrated to a dose equivalence to maintain at least 90% of hemodynamic response seen with the commerical product.
  In Part 2, subjects were treated with VentaProst only.
  Interventions: Combination Product: VentaProst

INTERVENTIONS:
Combination Product: VentaProst — epoprostenol for inhalation via custom drug delivery system

SUMMARY:
The purpose of the Phase 2a study is to: 1) demonstrate that the estimated VentaProst dose is safe and equivalent in effect to a dose administered via epoprostenol aerosolization by the current off-label-use practice; and 2) demonstrate that an optimum effect can be rapidly obtained with VentaProst titration.

DETAILED DESCRIPTION:
Part I:

This part of the study is designed to demonstrate the dose equivalence between off-label aerosolized epoprostenol and VentaProst using a patient's hemodynamic parameters.

Part II:

This part of the study is designed to establish a dose response relationship of VentaProst to hemodynamic effect by dose escalation in patients who have had cardiac surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

1. Women and Men 18 to 75 years of age
2. Provide written informed consent
3. Willing and able to comply with all aspects of the protocol
4. For patients in Part I:

   1. Undergo cardiac surgery on CPB
   2. Clinically require treatment with and receive aerosolized epoprostenol
   3. Demonstrate a clinically meaningful hemodynamic response to aerosolized epoprostenol
5. For patients in Part II:

   1. Undergo cardiac surgery with CPB
   2. Have perioperative pulmonary hypertension
   3. Clinically require treatment with inhaled epoprostenol

Exclusion Criteria:

1. Current smoker (i.e., within the last 30 days)
2. Emergency operative status
3. Upper and/or lower respiratory tract infection within four weeks of screening
4. Contraindication to transesophageal echocardiogram (TEE) including esophageal disease or unstable cervical spine
5. Renal or severe hepatic impairment
6. Thromboembolic disease treated with anticoagulant therapy
7. Bleeding disorders
8. Significant restrictive or obstructive lung disease
9. History of concurrent malignancy or recurrence of malignancy within two years prior to Screening
10. History of a diagnosis of drug or alcohol dependency or abuse within approximately the last three years
11. Recent history of stroke or transient ischemic attack
12. Significantly abnormal laboratory tests at Screening
13. Pregnant or breastfeeding
14. Treatment with an investigational drug, biologic, or device within 30 days
15. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator or Sponsor, would make the patient inappropriate for entry into this trial
16. Any condition where aerosolized epoprostenol is contraindicated
17. Known allergy or sensitivity to epoprostenol, any of its ingredients, or the diluent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hill, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University Medical Center, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- VentaProst: VentaProst (epoprostenol solution for inhalation via custom drug delivery system)
  VentaProst: Part I - an equivalent dose of VentaProst compared to conventionally-administered aerosolized epoprostenol with subsequent dose titration to achieve a clinically significant hemodynamic response Part II - Dose titration to achieve a clinically significant hemodynamic response.
Period: Part 1: Epoprostenol Then VentaProst
Arm/Group | VentaProst
Started | 9
Completed | 7
Not Completed | 2
Period: Part 2: VentaProst Dose Escalation
Arm/Group | VentaProst
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Epoprostenol Then VentaProst: an equivalent dose of VentaProst compared to conventionally-administered aerosolized epoprostenol with subsequent dose titration to achieve a clinically significant hemodynamic response
- Part 2: VentaProst Dose Escalation: Dose titration to achieve a clinically significant hemodynamic response.
- Total: Total of all reporting groups
Arm/Group | Part 1: Epoprostenol Then VentaProst | Part 2: VentaProst Dose Escalation | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (11.47) | 65.6 (8.02) | 65.8 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kg] | 85.6 (21.11) | 83.6 (17.57) | 84.5 (18.61)

OUTCOME MEASURES:

1. Primary Outcome: Identify Equivalent Dose of VentaProst Necessary to Achieve a PD Response Comparable to Standard of Care Treatment (Part I)
Description: The primary goal was to establish the dose of VentaProst necessary to achieve a PD response comparable to the standard of care. The first dose of VentaProst tested, 17 ng/kg/min, achieved the dose equivalency.
Time Frame: Pharmacodynamic changes will be measured during surgery (Day 1), post-surgery (Day 1), and from start of study treatment (Day 1) through study completion (up to 30 days)
Population: Per protocol population (Part I)
Measure: Number; unit: ng/kg/min
Arm/Group | VentaProst
Number analyzed (Participants) | 7
ng/kg/min | 17

2. Secondary Outcome: Optimal Dose Determination With VP Dose Escalation (Part II)
Description: Calculate vascular resistance indicators for CI and CO, and PAPi at each dose level. Identify the VP dose where mPAP, VR(CO), VR(CI), CVP are lowest, and CI/CO are highest. Compare in a narrative to the selected VP optimal dose by the Investigator by individual patient.
Time Frame: as for outcome 1
Population: Per protocol population (Part II)
Measure: Number; unit: ng/kg/min
Arm/Group | VentaProst
Number analyzed (Participants) | 8
ng/kg/min
  Optimal VP dose 1: number analyzed (Participants) | 2
  Optimal VP dose 1 | 6.8
  Optimal VP dose 2: number analyzed (Participants) | 3
  Optimal VP dose 2 | 10.2
  Optimal VP dose 3: number analyzed (Participants) | 3
  Optimal VP dose 3 | 13.6

ADVERSE EVENTS:
Time Frame: Adverse events were collect from post-cardiac surgery (Day 1) through study completion (up to 30 days).
Groups:
- Part 1: Epoprostenol Then VentaProst: an equivalent dose of VentaProst compared to conventionally-administered aerosolized epoprostenol
Arm/Group | Part 1: Epoprostenol Then VentaProst | Part 2: VentaProst Dose Escalation
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/8
Other Adverse Events (participants affected / at risk) | 2/7 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Epoprostenol Then VentaProst (N=7) | Part 2: VentaProst Dose Escalation (N=8)
pulmonary hypertension (Cardiac disorders) | 1 | 0
arterial hemorrhage (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Epoprostenol Then VentaProst (N=7) | Part 2: VentaProst Dose Escalation (N=8)
coagulopathy (Blood and lymphatic system disorders) | 1 | 0
adrenal insufficiency (Endocrine disorders) | 1 | 0
acute kidney injury (Renal and urinary disorders) | 1 | 0
acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0
traumatic hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
arterial hemorrhage (Vascular disorders) | 0 | 1
hemorrhage (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT03122730/Prot_SAP_000.pdf